CLINICAL TRIAL: NCT01756833
Title: Non-Invasive Treatment of Abdominal Aortic Aneurysm Clinical Trial (N-TA^3CT)
Brief Title: Non-Invasive Treatment of Abdominal Aortic Aneurysm Clinical Trial
Acronym: N-TA^3CT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Terrin, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00051170; R01AG037120 (NIH)
Record Dates: First submitted 2012-12-20; First posted 2012-12-28 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Aneurysm
Keywords: abdominal; aortic; aneurysm
MeSH Terms: conditions — Aneurysm | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Active Comparator): 100 mg capsules, twice a day, for a period of two years.
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): 100 mg capsules, twice a day, for a period of two years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — 100 mg po bid
  Other Names: doxycycline hyclate; Vibramycin; Oracea; Adoxa; Atridox and others
  Arms: Doxycycline
Drug: Placebo — capsule identical to the doxycycline capsule
  Other Names: capsule containing inert filler
  Arms: Placebo

SUMMARY:
The primary aim of this study is to determine if doxycycline (100 mg bid) will inhibit (by at least 40%) the increase in greatest transverse diameter of small abdominal aortic aneurysms (3.5-5.0 cm in men, 3.5-4.5 cm in women) over a 24-month period of observation in comparison to a placebo-treated control group.

DETAILED DESCRIPTION:
N-TA^3CT is a randomized, double-blind, placebo-controlled test of the hypothesis that doxycycline 100 mg bid, will reduce the rate of increase of maximum transverse diameter of small (3.5-5.0 cm among men and 3.5 to 4.5 cm among women) abdominal aortic aneurysms. The primary outcome is abdominal aortic aneurysm (AAA) maximum transverse diameter determined by CT scans at two-year follow-up with allowance for baseline (pre-randomization) diameter. Based on an anticipated growth rate of 2.5 mm per year in the placebo group and the current threshold at which surgical intervention will be offered to trial participants, (5.5 cm in men, 5.0 cm in women), the upper limit of AAA size for inclusion has been set at 5.0 cm for men and 4.5 cm for women. Among these subjects, the threshold for repair would be exceeded only by those exhibiting persistent growth. Secondary outcomes will determine if doxycycline affects other measures, e.g., MMP-9 levels in plasma and whether these effects are related to aneurysm growth. Nineteen clinical sites have identified pools of over 1600 patients with small aneurysm who meet the proposed inclusion/exclusion criteria. Two hundred fifty-eight patients will be randomized to placebo or doxycycline and their aneurysms followed for change in diameter at six-month intervals using CT imaging. The alternative hypothesis is that doxycycline will inhibit the expansion rate by 40% during the two years of observation. Patients enrolling in N-TA^3CT must be able to give consent for their participation themselves and meet study eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients 55 years of age or older, women post-surgical menopause or at least two years since last menses if natural menopause.
* CT scan documented infrarenal abdominal aortic aneurysm with maximum transverse diameter larger than 35 mm and no greater than 50 mm, in men, and larger than 35 mm and no greater than 45 mm in women.

Exclusion Criteria:

* Patients will be excluded from the study if they are unable to give their own informed consent to participate.
* have symptoms related to abdominal aortic aneurysm.
* have other intra-abdominal vascular pathology that may require repair within 24 months (e.g., renal artery stenosis, large iliac artery aneurysms, iliac occlusive disease, aneurysmal involvement of the renal artery).
* have had previous abdominal aortic aneurysm repair by open surgical or endovascular technique.
* have an active malignancy with life expectancy less than two years.
* have an allergy to tetracycline.
* are currently or have been recently treated (previous six months) with tetracycline derivatives.
* they are currently taking anti-seizure medicines metabolized by pathways influenced by doxycycline (e.g., carbamazepine, phenytoin, and barbiturates).
* stage II hypertension (patients whose blood pressure is persistently in the range of systolic > 160 mm Hg or diastolic > 100 mm Hg despite primary physician's best effort to achieve adequate therapy.
* have dialysis dependent renal failure or impending dialysis treatment for renal insufficiency.
* have a chronic infection requiring long-term (> 2 weeks) antibiotics.
* have known genetic syndromes responsible for the abdominal aortic aneurysm (e.g., Marfan's Syndrome).
* are under treatment with systemic immunosuppressive agents.
* could become pregnant.
* are not good candidates for clinical trial participation.
* are enrolled in another clinical trial.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Terrin, MD, Principal Investigator — University of Maryland, Baltimore; Bernard T Baxter, MD, Principal Investigator — University of Nebraska; Jonathan Matsumura, MD, Principal Investigator — University of Wisconsin Medical Center; John Curci, MD, Principal Investigator — Vanderbilt University
Locations (22):
- United States (22):
  - University of Arizona Medical Center, Tucson, Arizona
  - Carondelet Heart & Vascular Institute, Tucson, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Miami Cardiac and Vascular Institute, Miami, Florida
  - University of South Florida Health Center, Tampa, Florida
  - Northwestern University Memorial Hospital, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - McLaren Northern Michigan, Petoskey, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Omaha VAMC, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Portland VAMC, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Utah VAMC, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Baxter BT, Matsumura J, Curci J, McBride R, Blackwelder WC, Liu X, Larson L, Terrin ML; N-TA(3)CT Investigators. Non-invasive Treatment of Abdominal Aortic Aneurysm Clinical Trial (N-TA(3)CT): Design of a Phase IIb, placebo-controlled, double-blind, randomized clinical trial of doxycycline for the reduction of growth of small abdominal aortic aneurysm. Contemp Clin Trials. 2016 May;48:91-8. doi: 10.1016/j.cct.2016.03.008. Epub 2016 Mar 25. PMID 27018941
- [Background] Lachin JM. Worst-Rank Score Methods-A Nonparametric Approach to Informatively Missing Data. JAMA. 2020 Oct 27;324(16):1670-1671. doi: 10.1001/jama.2020.7709. No abstract available. PMID 32986071
- [Background] Lachin JM. Nonparametric Statistical Analysis. JAMA. 2020 May 26;323(20):2080-2081. doi: 10.1001/jama.2020.5874. No abstract available. PMID 32453350
- [Result] Baxter BT, Matsumura J, Curci JA, McBride R, Larson L, Blackwelder W, Lam D, Wijesinha M, Terrin M; N-TA3CT Investigators. Effect of Doxycycline on Aneurysm Growth Among Patients With Small Infrarenal Abdominal Aortic Aneurysms: A Randomized Clinical Trial. JAMA. 2020 May 26;323(20):2029-2038. doi: 10.1001/jama.2020.5230. PMID 32453369
- [Derived] Olson SL, Panthofer AM, Blackwelder W, Terrin ML, Curci JA, Baxter BT, Weaver FA, Matsumura JS; Non-Invasive Treatment of Abdominal Aortic Aneurysm Clinical Trial Investigators. Role of volume in small abdominal aortic aneurysm surveillance. J Vasc Surg. 2022 Apr;75(4):1260-1267.e3. doi: 10.1016/j.jvs.2021.09.046. Epub 2021 Oct 14. PMID 34655683
- [Derived] Panthofer AM, Olson SL, Rademacher BL, Grudzinski JK, Chaikof EL, Matsumura JS; N-TA(3)CT Investigators. Anatomic eligibility for endovascular aneurysm repair preserved over 2 years of surveillance. J Vasc Surg. 2021 Nov;74(5):1527-1536.e1. doi: 10.1016/j.jvs.2021.04.044. Epub 2021 May 4. PMID 33957227
- [Derived] Olson SL, Wijesinha MA, Panthofer AM, Blackwelder WC, Upchurch GR Jr, Terrin ML, Curci JA, Baxter BT, Matsumura JS. Evaluating Growth Patterns of Abdominal Aortic Aneurysm Diameter With Serial Computed Tomography Surveillance. JAMA Surg. 2021 Apr 1;156(4):363-370. doi: 10.1001/jamasurg.2020.7190. PMID 33595625

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxycycline | Placebo
Started | 133 | 128
Completed | 129 | 125
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: Seven participants who were randomized had insufficient follow-up to be included in the primary analysis. There were two patients whose baseline specimens were lost in shipment reducing the total number for baseline evaluations of MMP-9 and CRP from 254 to 252.
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Placebo | Total
Number analyzed (Participants) | 129 | 125 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (7.5) | 70.9 (7.3) | 71.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 111 | 108 | 219
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 122 | 119 | 241
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 3 | 4 | 7
  White | 120 | 113 | 233
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 129 | 125 | 254
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 44 | 43 | 87
  Former Smoker | 75 | 73 | 148
  Never Smoked | 10 | 9 | 19
Clinical History [Count of Participants; unit: Participants]
  Hypercholesterolemia | 98 | 98 | 196
  Coronary artery disease | 51 | 53 | 104
  Cancer | 44 | 38 | 82
  Chronic obstructive pulmonary disease | 30 | 29 | 59
  Diabetes | 35 | 22 | 57
  Family history of abdominal aortic aneurysm | 27 | 20 | 47
  Atrial fibrillation | 16 | 17 | 33
  Stroke | 13 | 15 | 28
  Congestive Heart Failure | 11 | 9 | 20
Medications [Count of Participants; unit: Participants]
  Statin | 104 | 103 | 207
  Any antihypertensive | 105 | 94 | 199
  B-Blocker | 68 | 63 | 131
  Diuretics | 43 | 40 | 83
  Angiotensin-converting enzyme inhibitor | 51 | 37 | 88
  Calcium channel blocker | 26 | 34 | 60
  Angiotensin receptor blocker | 20 | 25 | 45
  Aspirin or other antiplatelet | 95 | 92 | 187
  Daily aspirin | 86 | 89 | 175
  Other antiplatelet | 19 | 25 | 44
Aneurysm Diameter (Overall) [Mean (Standard Deviation); unit: cm] — Aneurysm values round to 4.3 cm (SD = 0.4 cm) for the total and for each of the two treatment groups.
  cm | 4.3 (0.4) | 4.3 (0.4) | 4.3 (0.4)
Aneurysm Diameter (Men) [Mean (Standard Deviation); unit: cm] — Population: Aneurysm diameter (cm) measured in men
  cm
    number analyzed (Participants) | 111 | 108 | 219
    (all) | 4.3 (0.4) | 4.4 (0.4) | 4.4 (0.4)
Aneurysm Diameter (Women) [Mean (Standard Deviation); unit: cm] — Population: Aneurysm diameter (cm) measured in women
  cm
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 4.1 (0.3) | 3.9 (0.3) | 4.0 (0.3)
Aneurysm Volume (Overall) [Mean (Standard Deviation); unit: cm^3] | 97.0 (24.0) | 95.8 (24.0) | 96.4 (24.0)
Aneurysm Volume (Men) [Mean (Standard Deviation); unit: cm^3] — Population: Aneurysm volume (cm3) measured in men
  cm^3
    number analyzed (Participants) | 111 | 108 | 219
    (all) | 99.0 (24.3) | 99.2 (23.3) | 99.1 (23.8)
Aneurysm Volume (Women) [Mean (Standard Deviation); unit: cm^3] — Population: Aneurysm volume (cm3) measured in women
  cm^3
    number analyzed (Participants) | 18 | 17 | 35
    (all) | 84.9 (18.5) | 74.3 (15.9) | 79.6 (16.7)
MMP-9 Levels (ng/ml) [Mean (Standard Deviation); unit: ng/ml] — Population: MMP-9 levels (ng/ml) measured at baseline
  ng/ml
    number analyzed (Participants) | 128 | 124 | 252
    (all) | 54.6 (53.2) | 55.0 (51.1) | 54.8 (52.1)
CRP Levels, mg/l [Mean (Standard Deviation); unit: mg/l] — Population: CRP Levels (mg/l) measured at baseline
  mg/l
    number analyzed (Participants) | 128 | 124 | 252
    (all) | 5.4 (13.6) | 3.6 (4.9) | 4.5 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Z-score for Rank of Maximum Transverse Diameter (MTD) Regressed on Z-score at Baseline to Assess Growth in Abdominal Aortic Aneurysm MTD Determined by CT Scans at Two-year Follow-up and Baseline (Pre-randomization).
Description: Diameters were ranked from smallest to largest. Worse ranks were assigned to surviving patients who underwent aneurysm repair (in order of longest to shortest time from randomization to repair), and worst ranks were assigned to patients who died (in order likewise). Each rank was converted to a z-score corresponding to the value on the standard normal curve of its percentile. The primary analysis was based on linear regression of the change in z-scores from baseline to 2 years. Independent variables were baseline z-score, sex, and a dichotomous variable for the randomly assigned treatment group (0 for placebo, 1 for doxycycline). Missing values were multiply imputed. Higher score corresponds to less favorable outcome. There is no scale associated with these z-scores; the absolute z-scores have no biological meaning or clinically relevant threshold. A z-score of 0 corresponds to the median rank. The maximum and minimum z-scores are +2.41 and -2.41. See References in Protocol Section.
Time Frame: Baseline and two years from randomization (when patients were late in returning for visits, their data were used up to three years).
Population: The number of participants refers to the number for whom CT scans were available.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
z-score | 0.0262 (1.0) | -0.0258 (1.0)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; Null hypothesis: normal score of MTD at follow-up adjusted for baseline and gender in doxycycline assigned patients - normal score of MTD at follow-up adjusted for baseline and gender in placebo assigned patients = 0. Sample size: The criterion ("alpha") set for statistical significance was 1-sided .025; use of this level means that the inference from the test result will be the same as the inference from 2-sided testing at the .05 significance level; Test type: Superiority; p = 0.71, ANCOVA on normal scores — Two prespecified interim analyses for efficacy performed when 1/3 & 2/3 of primary outcome available, significance level, 1-sided, alpha=.0005. Final analysis 1-sided, alpha=.024. Futility analysis performed when ~2/3 primary outcome was available; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.07 to 0.07], Standard Deviation 0.035; For the primary analysis, diameters at baseline were ranked from smallest to largest (ranks 1-254). At the 2-year follow-up, ranks 1 through 225 were assigned to the diameters of surviving patients with no aneurysm repair (with missing values estimated by multiple imputation), ranks 226 through 247 were assigned to surviving patients who underwent aneurysm repair (in order of longest to shortest time from randomization to repair), and ranks 248 through 254 were assigned to patients who died (in order of longest to shortest time from randomization to death). Each rank was converted to a normal score corresponding to the value on the standard normal curve (z score) of its percentile among all 254 ranks. The primary analysis was based on linear regression of the change in normal scores from baseline to 2 years. Independent variables were baseline normal score, sex, and a dichotomous variable for the randomly assigned treatment group (0 for placebo, 1 for doxycycline)

2. Secondary Outcome: Maximum Transverse Diameter, cm
Description: Secondary outcomes will derive from central, Imaging Core Laboratory analyses of the CT scans performed every six months on patients and from the clinical follow-up of randomized patients, from clinical observation, local laboratory findings, study visit quality of life assessments, and from biomarker analyses to be performed in the Biomarkers Core Laboratory (e.g., changes from initial matrix metalloproteinase (MMP-9) levels, and matrix metalloproteinase (MMP-9) levels at 24 months). When patients were late in returning for visits their data were used up to three years.
Time Frame: Six months, one year, and two years (when patients were late in returning for visits their data were used up to three years).
Population: All patients for whom any follow-up CT scans of the abdomen and pelvis were obtained.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
cm
  Maximum Transverse Diameter, cm 6 months: number analyzed (Participants) | 119 | 116
  Maximum Transverse Diameter, cm 6 months | 4.40 (0.44) | 4.40 (0.43)
  Maximum Transverse Diameter, cm 1 year: number analyzed (Participants) | 119 | 113
  Maximum Transverse Diameter, cm 1 year | 4.49 (0.48) | 4.48 (0.44)
  Maximum Transverse Diameter, cm 2 year: number analyzed (Participants) | 96 | 101
  Maximum Transverse Diameter, cm 2 year | 4.61 (0.52) | 4.61 (0.53)
  Maximum Transverse Diameter, cm Baseline to 2 year change: number analyzed (Participants) | 96 | 101
  Maximum Transverse Diameter, cm Baseline to 2 year change | 0.36 (0.21) | 0.36 (0.28)

3. Secondary Outcome: Volume, cm^3
Description: as for outcome 2
Time Frame: as for outcome 2
Population: All patients for whom any follow-up CT scans of the abdomen and pelvis were obtained.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
cm^3
  Volume, cm^3 6 months: number analyzed (Participants) | 119 | 116
  Volume, cm^3 6 months | 102.90 (26.19) | 100.40 (26.27)
  Volume, cm^3 1 year: number analyzed (Participants) | 119 | 113
  Volume, cm^3 1 year | 106.00 (29.13) | 105.00 (28.28)
  Volume, cm^3 2 year: number analyzed (Participants) | 96 | 101
  Volume, cm^3 2 year | 113.60 (34.91) | 111.20 (33.14)
  Volume, cm^3 Baseline to 2 year change: number analyzed (Participants) | 96 | 101
  Volume, cm^3 Baseline to 2 year change | 18.60 (14.38) | 19.16 (15.75)

4. Secondary Outcome: MMP-9, ng/ml
Description: Secondary outcomes will derive from central, Imaging Core Laboratory analyses of the CT scans performed every six months on patients and from the clinical follow-up of randomized patients, from clinical observation, local laboratory findings, study visit quality of life assessments, and from biomarker analyses to be performed in the Biomarkers Core Laboratory (e.g., changes from initial matrix metalloproteinase (MMP-9) levels, and matrix metalloproteinase (MMP-9) levels at 24 months). When patients were late in returning for visits their data were used up to three years.
  Analysis of hs-CRP will be performed using an immunoturbidimetric latex agglutination method (K-assay [KAI-60], Kamiya Biomedical Co., Seattle, WA).
Time Frame: Six months, one year, 18 months, and two years (when patients were late in returning for visits their data were used up to three years).
Population: All patients for whom any follow-up CT scans of the abdomen and pelvis were obtained.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
ng/ml
  MMP-9, ng/ml 6 months: number analyzed (Participants) | 108 | 111
  MMP-9, ng/ml 6 months | 60.9 (85.3) | 61.9 (61.8)
  MMP-9, ng/ml 1 year: number analyzed (Participants) | 111 | 100
  MMP-9, ng/ml 1 year | 63.0 (90.1) | 61.0 (91.5)
  MMP-9, ng/ml 1 year, 6 months: number analyzed (Participants) | 88 | 89
  MMP-9, ng/ml 1 year, 6 months | 48.8 (43.9) | 68.3 (86.7)
  MMP-9, ng/ml 2 year: number analyzed (Participants) | 86 | 83
  MMP-9, ng/ml 2 year | 53.8 (54.8) | 52.8 (41.9)

5. Secondary Outcome: CRP, mg/l
Description: Secondary outcomes will derive from central, Imaging Core Laboratory analyses of the CT scans performed every six months on patients and from the clinical follow-up of randomized patients, from clinical observation, local laboratory findings, study visit quality of life assessments, and from biomarker analyses to be performed in the Biomarkers Core Laboratory (e.g., changes from initial matrix metalloproteinase (MMP-9) levels, and matrix metalloproteinase (MMP-9) levels at 24 months). When patients were late in returning for visits their data were used up to three years.
  Plasma MMP-9 concentrations will be measured by an ELISA, two-site sandwich method that is commercially available (R & D Systems, Quantikine, DMP900).
Time Frame: as for outcome 4
Population: All patients for whom any follow-up CT scans of the abdomen and pelvis were obtained.
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
mg/l
  CRP, mg/l 6 months: number analyzed (Participants) | 108 | 111
  CRP, mg/l 6 months | 5.4 (12.7) | 4.5 (10.7)
  CRP, mg/l 1 year: number analyzed (Participants) | 111 | 100
  CRP, mg/l 1 year | 3.5 (4.8) | 4.1 (6.9)
  CRP, mg/l 1 year, 6 months: number analyzed (Participants) | 88 | 89
  CRP, mg/l 1 year, 6 months | 3.5 (6.5) | 5.7 (15.1)
  CRP, mg/l 2 year: number analyzed (Participants) | 86 | 83
  CRP, mg/l 2 year | 5.9 (15.6) | 4.0 (5.3)

6. Other Pre Specified Outcome: Number of Participants With Aneurysm Rupture
Description: Clinically reported rupture events.
Time Frame: Two years
Population: Full analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
Participants | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Surgical Intervention
Description: Clinically reported aneurysm repair.
Time Frame: Two years
Population: Full analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
Participants | 13 | 9

8. Other Pre Specified Outcome: Number of Participants Who Died
Description: Clinically reported deaths.
Time Frame: Two years
Population: Full analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 129 | 125
Participants | 3 | 4

ADVERSE EVENTS:
Time Frame: Two years
Description: Adverse Events were classified without regard to specific Adverse Event Term.
Arm/Group | Doxycycline | Placebo
All-Cause Mortality (participants affected / at risk) | 3/129 | 4/125
Serious Adverse Events (participants affected / at risk) | 70/129 | 71/125
Other Adverse Events (participants affected / at risk) | 121/129 | 111/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (N=129) | Placebo (N=125)
Serious or Unexpected Adverse Events (Cardiac disorders) | 14 (18) | 11 (16)
Serious or Unexpected Adverse Events (Gastrointestinal disorders) | 14 (27) | 16 (24)
Serious or Unexpected Adverse Events (General disorders) | 10 (13) | 11 (18)
Serious or Unexpected Adverse Events (Infections and infestations) | 12 (15) | 6 (6)
Serious or Unexpected Adverse Events (Injury, poisoning and procedural complications) | 6 (9) | 7 (10)
Serious or Unexpected Adverse Events (Metabolism and nutrition disorders) | 4 (4) | 2 (6)
Serious or Unexpected Adverse Events (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (11)
Serious or Unexpected Adverse Events (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (9) | 6 (6)
Serious or Unexpected Adverse Events (Nervous system disorders) | 10 (21) | 6 (8)
Serious or Unexpected Adverse Events (Renal and urinary disorders) | 5 (9) | 6 (6)
Serious or Unexpected Adverse Events (Respiratory, thoracic and mediastinal disorders) | 12 (23) | 12 (22)
Serious or Unexpected Adverse Events (Surgical and medical procedures) | 32 (36) | 38 (45)
Serious or Unexpected Adverse Events (Vascular disorders) | 5 (7) | 7 (8)
Serious or Unexpected Adverse Events (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Serious or Unexpected Adverse Events (Psychiatric disorders) | 3 (3) | 2 (2)
Serious or Unexpected Adverse Events (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Serious or Unexpected Adverse Events (Social circumstances) | 1 (1) | 0 (0)
Serious or Unexpected Adverse Events (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Serious or Unexpected Adverse Events (Endocrine disorders) | 0 (0) | 1 (1)
Serious or Unexpected Adverse Events (Eye disorders) | 1 (1) | 0 (0)
Serious or Unexpected Adverse Events (Hepatobiliary disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxycycline (N=129) | Placebo (N=125)
Frequent joint pain (Musculoskeletal and connective tissue disorders) | 84 (84) | 79 (79)
Frequent gastric or intestinal upset (Gastrointestinal disorders) | 58 (58) | 56 (56)
Frequent bleeding or bruising (Blood and lymphatic system disorders) | 47 (47) | 54 (54)
Frequent spells of dizziness (General disorders) | 34 (34) | 37 (37)
Skin rash or hives (Skin and subcutaneous tissue disorders) | 41 (41) | 29 (29)
Visual disturbance (Eye disorders) | 26 (26) | 43 (43)
Moderate to severe sunburn (Skin and subcutaneous tissue disorders) | 38 (38) | 14 (14)
Frequent headaches (General disorders) | 27 (27) | 20 (20)
Tooth discoloration (General disorders) | 12 (12) | 18 (18)
Fever (General disorders) | 11 (11) | 18 (18)
Other symptom requiring study drug dose adjustment or discontinuation (General disorders) | 27 (27) | 27 (27)

LIMITATIONS AND CAVEATS:
Follow-up was limited to two years for most patients and results could differ with longer term follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-04-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT01756833/Prot_003.pdf
  • Statistical Analysis Plan (2017-03-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT01756833/SAP_001.pdf
  • Informed Consent Form (2015-02-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT01756833/ICF_004.pdf